CLINICAL TRIAL: NCT04400006
Title: The Effectiveness of Ozone Therapy in the Prevention of COVID-19 Infection
Brief Title: Ozone Therapy in the Prevention of COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Kardelen Gencer Atalay, Principal Investigator, Marmara University
Other Study IDs: 2761
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Corona Virus Infection
Keywords: Coronavirus; Ozone; Preventive Medicine
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus has already infected 4,673,809 people and killed 312,646 people worldwide, and no specific treatment or a vaccine against it has yet proven to be effective. Ozone therapy has become o promising tool for both prevention and treatment of COVID-19 infection by various possible mechanisms. The oxidative stress created by ozone in the body to stimulate the peripheral phagocytic cells, activate the antioxidant system, and restore the immune system is thought to be effective for the prevention of COVID-19 infection.

In recent years, ozone therapy has become a popular alternative method for chronic pain management of various diseases such as fibromyalgia, knee osteoarthritis, and rheumatic diseases. As a result of this, there were many individuals who had received ozone therapy before the outbreak of COVID-19. This study aimed to investigate the preventive effect of ozone therapy against COVID-19 infection in these individuals.

DETAILED DESCRIPTION:
The inclusion criteria were determined to be completed at least ten sessions of ozone therapy applied by the method of major autohemotherapy in the last six months from the time the first COVID-19 case of Turkey reported (Mar 11, 2020). Individuals who received ozone therapy locally or fewer than ten sessions, who did not want to participate were excluded.

The major autohemotherapy procedure to all the participants was applied as follows: 100mL of blood was drawn by a vacuum from the antecubital vein into a sterile glass bottle in which 12 mL of 3.13% sodium citrate solution as an anticoagulant (MediPac®, Germany). A corresponding volume (100mL) of gas with an ozone concentration of 10-20 µg/mL was immediately added and continuously mixed by a gentle rotating movement to avoid foaming to the blood in the bottle. Ozone was produced by a Blue-S medical ozone generator (Turkozone®, Turkey). Reinfusion was accomplished in about 15-20 minutes, and the whole procedure was carried out in approximately 30 minutes and was repeated two or three times a week.

ELIGIBILITY:
Inclusion Criteria:

* To be completed at least ten sessions of ozone therapy applied by the method of major autohemotherapy in the last six months from the time the first COVID-19 case of Turkey reported (Mar 11, 2020)

Exclusion Criteria:

* To received ozone therapy locally or fewer than ten sessions
* not want to participate

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals who completed at least ten sessions of ozone therapy applied by the method of major autohemotherapy* in the last six months from the time the first COVID-19 case of Turkey reported (Mar 11, 2020).
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
The survey that was taken by telephone calls | Day 0
  It involved questions about age, gender, height, weight, occupation, comorbidities, and concurrent medications, in addition to a detailed query for COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Kardelen Gencer, Principal Investigator — Marmara University
Locations (1):
- Kardelen Gencer Atalay, Istanbul, Turkey (Türkiye)